CLINICAL TRIAL: NCT05374109
Title: SYV: A Mental Health Intervention to Improve HIV Outcomes in Tanzanian Youth
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Kilimanjaro Christian Medical Centre, Tanzania (Other); National Institute for Medical Research, Tanzania (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00109309; 1R01MH124476-01A1 (NIH)
Record Dates: First submitted 2022-05-06; First posted 2022-05-16 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: HIV-1-infection; Mental Health Issue; Adherence, Medication
Keywords: HIV-1; Adolescent; Youth; Mental Health; Africa; Tanzania; Medication Adherence
MeSH Terms: conditions — Medication Adherence; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Restricted randomization will be used to balance the randomization across both study arms by site, sex, and enrollment HIV RNA (<400 copies/mL or ≥400 copies/mL). Those randomized to receive the SYV intervention will be assembled into 33 groups of 10-11 participants per group. Those randomized to SOC will continue to receive routine care, which will be clearly defined by each site. The outcomes assessor and statisticians will be masked to participant study arm through the 6-month study visit (primary aim).
Who Masked: Outcomes Assessor
Masking Description: The research assistant asking participants questions and the statistician are masked (not aware to which group participants were randomized).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SYV: Sauti ya Vijana (The Voice of Youth intervention) (Active Comparator): Sessions 1 to 3 - youth name their worries, discuss coping strategies, practice relaxation and breathing exercises, and learn components of cognitive behavioral therapy. Sessions 4 to 6 are dedicated to reflection and processing trauma. Caregivers (supportive adults) are invited at the discretion of enrolled youth to participate in Sessions 1 and 6. Session 7 - youth name their support network and any changes. Sessions 8 and 9 - youth consider stigma, disclosure, reproductive health, condom use, and gender-based violence. Sessions 9 and 10 expand the overall client-centered approach to emphasizing autonomy rather than imposing ideas about what the youth "should" do. In a final individual meeting, youth revisit their personal values, goals, and strategies for the next 6 months and review their support networks. A final gathering is used to review all session content, to celebrate all that has been shared and learned together, and to distribute certificates of completion.
  Interventions: Behavioral: SYV: Sauti ya Vijana (The Voice of Youth intervention)
- SOC - Standard of Care (No Intervention): Participants in the SOC will not meet in study groups, thus are more "at risk" for attrition. They will be contacted by the study team on a monthly basis to check in and ensure their documented contact information remains accurate. SOC may vary by site depending on clinic structure, referral systems, and group activities. These differences could potentially dilute the SYV intervention effect and introduce content spillover whereby participants randomized to the intervention discuss intervention content with participants randomized to SOC. As part of the study survey, participants will be asked if they had friends who attended the SYV intervention and if they discussed content. Additionally, as part of the implementation science outcomes (Aim 3), the SOC group structure, adherence counseling, and any mental health referrals offered as part of SOC will be documented.

INTERVENTIONS:
Behavioral: SYV: Sauti ya Vijana (The Voice of Youth intervention) — Mental health is associated with ART adherence and HIV outcomes. SYV was designed to address the specific challenges of young people living (YPLWH) with HIV in Tanzania. SYV includes 10 group sessions (two sessions held jointly with caregivers) lasting approximately 90 minutes and two individual sessions delivered by trained young adult group leaders who use a manualized protocol that is designed to scale in low resource settings. The intervention is applied to the Social Action Theory (SAT), a theoretical framework used to determine factors that influence health behavior. Building off a SAT resilience framework for YPLWH, components of evidence-based treatment models to influence cognitive, self, and social regulation to improve behavioral health outcomes will be strategically used.
  Arms: SYV: Sauti ya Vijana (The Voice of Youth intervention)

SUMMARY:
The overall objectives of this proposal are to support positive coping strategies that bolster mental health and lead to improved HIV outcomes among Young People Living with HIV (YPLWH). The central hypothesis is that SYV (Sauti ya Vijana, The Voice of Youth) will be effective to improve antiretroviral therapy (ART) adherence and virologic suppression in YPLWH in Tanzania. The rationale for this project is that by targeting mental health, which is strongly associated with medication adherence, that this will effectively improve adherence and thereby HIV viral suppression. The central hypothesis will be tested in three aims in a hybrid type-1 effectiveness-implementation trial.

DETAILED DESCRIPTION:
The rigorous experimental design includes a pilot study followed by a parallel-arm randomized control trial (RCT). The pilot will include approximately eight consenting members of the youth community advisory board (CAB) at each site location prior to the RCT. If a youth CAB does not currently exist at each site, one will be formed. Although the investigators have strong pilot data for the SYV intervention from Moshi, the pilot test proposed herein will help ensure recruitment, enrollment, intervention delivery, supervision, measurement technology and logistics run as expected at each site (Moshi, Mbeya, Mwanza, Ifakara). The pilot study will be comprised of 8 participants recruited at each site. Subsequently, for the RCT, we will individually randomize up to 750 participants to receive the SYV intervention or SOC (standard of care) to achieve 90% power to detect a 10 percentage point difference between arms in the primary outcome of virologic suppression at the two-tailed 5% significance level, accounting for clustering by SYV group in the intervention arm.

The intervention will be rolled out across four main sites, in four different Tanzanian regions, and in four waves separated in time by 6 months. There will be two SYV groups per wave at each site (~8 groups per site) A study visit for all participants will be conducted baseline and approximately 4 months (T1), 6-, 12-, and 18-months post-baseline (T2, T3, T4) with 6-months post baseline being the primary endpoint. At 12 months post-baseline (T3), those randomized to the SYV intervention will receive a one-session SYV booster to improve content retention and study engagement as has been shown in prior studies.

ELIGIBILITY:
Inclusion Criteria:

* Youth between the ages of 10 and 24 years of age
* Attending the enrolling adolescent HIV clinic
* Are fully disclosed and aware of their HIV status
* Receiving ART for a minimum of 6 months
* If ≥ 18 years, able to understand the project and provide written informed consent
* If <18 years, a parent or guardian must provide written permission and participant must be able to assent
* All adolescents must also commit to attending the 10 weekly SYV sessions and 2 individual sessions

Exclusion Criteria:

* Active psychosis
* Developmental delay, or cognitive disability that precludes active participation in consent process, intervention, and assessment interviews

Ages: 10 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 690 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-01-11 (Actual); Study Completion 2026-01-06 (Estimated)

PRIMARY OUTCOMES:
Virologic suppression as measured by percent of patients with a HIV RNA <400 copies/mL | 6 months post-baseline visit
  HIV RNA measured by blood testing

SECONDARY OUTCOMES:
Change in virologic suppression as measured by percent of patients with a HIV RNA <400 copies/mL | Baseline, months 4 and 12 post-baseline visit
  HIV RNA measured by blood testing
Change in virologic suppression as measured by percent of patients with a HIV RNA <200 copies/mL | Baseline, months 4, 6 and 12 post-baseline visit
  HIV RNA measured by blood testing
Change in virologic suppression as measured by percent of patients with a HIV RNA <50 copies/mL | Baseline, months 4, 6 and 12 post-baseline visit
  HIV RNA measured by blood testing
Change in HIV RNA log scale | Baseline, months 4, 6 and12 post-baseline visit in SYV intervention compared to standard of care.
  HIV RNA measured by blood testing
Change in the percentage of patients who are HIV RNA undetectable (<400 copies m/L) as measured by blood test | Baseline, months 4, 6, 12 and 18 post-baseline visit
  HIV RNA results
Change in the percentage of patients who are HIV RNA detectable (>400 copies m/L) as measured by blood test | Baseline, months 4, 6, 12 and 18 post-baseline visit
  HIV RNA results
Change in anti-retroviral therapy (ART) adherence as measured by SYV (Sauti ya Vijana) Scale - Adherence section | Baseline, months 4, 6, 12 and 18 post-baseline visit
  SYV Scale - Adherence section (Likert scale - not applicable)
Change in anti-retroviral therapy (ART) adherence as measured by concentration of ART medication(s) in hair sample | Baseline, months 4, 6, 12 and 18 post-baseline visit
  hair samples sent for analysis
Change in mental health status as measured by SYV Scale - General Anxiety Disorder-7 (GAD-7) section | Baseline, 4, 6, 12 and 18 months post-baseline visit
  SYV Scale - General Anxiety Disorder-7 (GAD-7) section (Likert scale 0 not at all to 3 nearly every day) 0 is the most positive choice
Change in mental health status as measured by SYV Scale - Patient Health Questionnaire-9 (PHQ-9) section | Baseline, 4, 6, 12 and 18 months post-baseline visit
  SYV Scale - Patient Health Questionnaire-9 (PHQ-9) section (Likert scale 0 not at all to 3 nearly every day) 0 is the most positive choice
Change in mental health status as measured by SYV Scale - Strengths and Difficulties Questionnaire (SDQ) section | Baseline, 4, 6, 12 and 18 months post-baseline visit
  SYV Scale - Strengths and Difficulties Questionnaire (SDQ) section (Likert scale 0 never true of me to 2 usually true of me) 0 or 2 can be most positive or most negative choices depending on the question
Change in mental health status as measured by SYV Scale - Self-Esteem section | Baseline, 4, 6, 12 and 18 months post-baseline visit
  SYV Scale - Self-Esteem section (Likert scale - 4 options from strongly agree to strongly disagree - no choice is most positive)
Change in mental health status as measured by SYV Scale - Adverse Childhood Experiences International Questionnaire (ACE-IQ) section | Baseline, 4, 6, 12 and 18 months post-baseline visit
  SYV Scale - Adverse Childhood Experiences International Questionnaire (ACE-IQ) section (Likert scale - 5 options from Always to Never - Always is the most positive choice, 5 options Many Times, A few times, Once, Never or Refused - Never is the most positive choice, 4 options None, Little, Much and Most - no choice is the most positive and 3 options are Yes, No or Not Sure - No is the most positive choice)
Change in coping habits as measured by SYV Scale - Adverse Childhood Experiences International Questionnaire (ACE-IQ) section | Baseline, 4, 6, 12 and 18 months post-baseline visit
  SYV Scale - Adverse Childhood Experiences International Questionnaire (ACE-IQ) section (Likert scale - 5 options from Always to Never - Never is the most positive choice, 5 options Many Times, A few times, Once, Never or Refused - Never is the most positive choice, 4 options None, Little, Much and Most - no choice is most positive and 3 options are Yes, No or Not Sure - No is the most positive choice)
Change in resilience as measured by SYV Scale - Adapted People Living with HIV Resilience Scale | Baseline, 4, 6, 12 and 18 months post-baseline visit
  SYV Scale - Adapted People Living with HIV Resilience Scale (Likert scale 5 options from strongly disagree to strongly agree - strongly agree is the most positive choice)
Change in stigma as measured by SYV Scale - Stigma section | Baseline, 4, 6, 12 and 18 months post-baseline visit
  SYV Scale - Stigma section (Likert scale 1 strongly disagree to 4 strongly agree - no most positive choice)
Change in overall quality of life measured by SYV Scale - Quality of Life (QOL) | Baseline, 4, 6, 12 and 18 months post-baseline visit
  SYV Scale - Quality of Life (QOL) (Likert scale 5 options from very poor/very dissatisfied to very good/very satisfied - very good/very satisfied is the most positive choice)
Change in gender based violence as measured by SYV Scale - Violence against partner section | Baseline, 4, 6, 12 and 18 months post-baseline visit
  SYV Scale - Violence against partner section (Likert scale Yes or No - No is the most positive choice)
Change in gender based violence as measured by SYV Scale - Violence Perpetration section | Baseline, 4, 6, 12 and 18 months post-baseline visit
  SYV Scale - Violence Perpetration section (Likert scale Yes or No - No is the most positive choice)
Change in disclosure as measured by SYV Scale - Stigma section | Baseline, 4, 6, 12 and 18 months post-baseline visit
  SYV Scale - Stigma section (Likert scale 1 strongly disagree to 4 strongly agree - strongly disagree is the most positive choice) and Sexual section (Likert scale - N/A)
Change in HIV knowledge as measured by SYV Scale - HIV Knowledge Questionnaire-18 (HIV-KQ-18) section | Baseline, 4, 6, 12 and 18 months post-baseline visit
  SYV Scale - HIV Knowledge Questionnaire-18 (HIV-KQ-18) section (Likert scale True/False/I don't know - no most positive choice)
Change in sexual high-risk behaviors as measured by SYV Scale - Sexual section | Baseline, 4, 6, 12 and 18 months post-baseline visit
  SYV Scale - Sexual section (Likert scale - N/A)
Change in substance abuse high-risk behaviors as measured by SYV Scale - Personal section | Baseline, 4, 6, 12 and 18 months post-baseline visit
  SYV Scale - Personal section (Likert scale N/A)

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy E Dow, MD, Principal Investigator — Duke University
Locations (6):
- Tanzania (6):
  - Chronic Disease Clinic of Ifakara Health Institute, Ifakara
  - Baylor College of Medicine Children's Foundation - Tanzania, Mbeya Centre for Excellence, Mbeya
  - Kilimanjaro Christian Medical Centre, Moshi
  - Mawenzi Regional Referral Hospital, Moshi
  - Baylor College of Medicine Children's Foundation - Tanzania, Mwanza Centre for Excellence, Mwanza
  - Bugando Medical Centre, Mwanza

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be de-identified and deposited in data repository alongside supporting documentation including but not limited to: readme file(s), blank data collection instruments, codebook(s), and/or data management program code. Additionally, analytic datasets and associated code may be deposited in conjunction with publications to facilitate replication of results.
  The data repository will be UNC Dataverse and the deposit will be part of the Adolescent Mental Health in Africa Network Initiative (AMANI) Dataverse (subject to change). A data curator will review the dataset prior to deposit in a repository to assess deductive disclosure risk. Terms of Use, a data use agreement, or other access restrictions may be implemented if limited access is determined appropriate for this study data; otherwise the data deposit within the repository will be open access.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: All collected IPD will be deposited in a repository within one year of the study's completion. It may be embargoed with the repository for a period of time to allow the study team to publish. Analytic datasets related to specific publications will be shared within one year of the publication date.
Access Criteria: The mechanism for sharing data is deposit in a data repository. Terms of Use, a data use agreement, or other access restrictions may be implemented if limited access is determined appropriate for this study data; otherwise the data deposit within the repository will be open access. If any access restrictions apply, the study PI will be responsible for reviewing and approving requests by other researchers to access the data. Other researchers may use published data for purposes allowed under applicable Terms of Use, data use agreements, and any other relevant policy, regulatory or legal restrictions.

REFERENCES:
- [Background] Dow DE, Mmbaga BT, Gallis JA, Turner EL, Gandhi M, Cunningham CK, O'Donnell KE. A group-based mental health intervention for young people living with HIV in Tanzania: results of a pilot individually randomized group treatment trial. BMC Public Health. 2020 Sep 4;20(1):1358. doi: 10.1186/s12889-020-09380-3. PMID 32887558
- [Background] Dow DE, Mmbaga BT, Turner EL, Gallis JA, Tabb ZJ, Cunningham CK, O'Donnell KE. Building resilience: a mental health intervention for Tanzanian youth living with HIV. AIDS Care. 2018;30(sup4):12-20. doi: 10.1080/09540121.2018.1527008. Epub 2019 Jan 9. PMID 30626197
- [Background] Mollel GJ, Ketang'enyi E, Komba L, Mmbaga BT, Shayo AM, Boshe J, Knettel B, Gallis JA, Turner EL, O'Donnell K, Baumgartner JN, Ogbuoji O, Dow DE. Study protocol for Sauti ya Vijana (The Voice of Youth): A hybrid-type 1 randomized trial to evaluate effectiveness and implementation of a mental health and life skills intervention to improve health outcomes for Tanzanian youth living with HIV. PLoS One. 2024 Aug 26;19(8):e0305471. doi: 10.1371/journal.pone.0305471. eCollection 2024. PMID 39186768
- [Background] Zimmerman A, Fawole A, Shahid M, Dow D, Ogbuoji O. Evidence Gaps in Economic Evaluations of HIV Interventions Targeting Young People: A Systematic Review. J Adolesc Health. 2024 Nov;75(5):709-724. doi: 10.1016/j.jadohealth.2024.06.013. Epub 2024 Aug 13. PMID 39140926
- See also: website with information regarding Sauti ya Vijana (The Voice of Youth) — http://sites.duke.edu/sautiyavijana

DOCUMENTS (1):
  • Informed Consent Form (2022-08-03): https://cdn.clinicaltrials.gov/large-docs/09/NCT05374109/ICF_000.pdf